CLINICAL TRIAL: NCT03467022
Title: Alcohol Abuse or Alcohol Withdrawal: Risk of Latent Scurvy: A STROBE Compliant Study
Brief Title: Alcohol Abuse or Alcohol Withdrawal: Risk of Latent Scurvy
Status: Completed | Type: Observational
Sponsor: SCP Battistelli (Other)
Responsible Party: Principal Investigator, Daniel Battistelli, Director, SCP Battistelli
Other Study IDs: SCPBattistelli
Record Dates: First submitted 2018-01-18; First posted 2018-03-15 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Alcoholics
Keywords: alcohol withdrawal; scurvy; vitamin C; tiredness
MeSH Terms: conditions — Scurvy; Fatigue | interventions — Ascorbic Acid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Measurement of vitamin C ail be performed by high-pressure liquid chromatography (Cerba Laboratory, F-Cergy Pontoise).
  Results are expressed in micromol per liter (µmol/L) with a normal range from 26,4 to 84,0µmol/L. These measures are in correlation with those quoted by O.Frain et al concerning healthy French men and women (5 to 15 mg/L equal to 28,4 -85,5µmol/L). According to Johnston's criteria, plasma vitamin C level lower than 11,4µmol/L (2mg/L) will be considered as vitamin C deficiency, lower than 28,4µmol/L (5 mg/L) as vitamin C depletion. The lower limit of quantification is 3µmol/L (< 0,5 mg /L); the patient is considered biologically as having scurvy or at high risk for development of scurvy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vitamin C — Patients depleted or deficient in vitamin C by blood test were supplemented orally in vitamin C 1 gram per day for three months
  Other Names: Ascorbic acid

SUMMARY:
Scurvy, or latent scurvy, may be underestimated in developed countries, but continue to be described, often as case report. Little is known about the prevalence of vitamin C deficiency in a specific population as withdrawal alcoholics and about his possible consequences, latent scurvy.

In an observational study, the investigators will evaluate prospectively the prevalence of vitamin C deficiency in alcoholic withdrawal patients, its correlation with latent scurvy, mainly tiredness and weakness, and the evolution of the latter at three months after oral vitamin C supplementation.

DETAILED DESCRIPTION:
This study aims to examine:

1. the level of plasma vitamin C for patients that volunteered for alcohol withdrawal. Measurement of vitamin C plasma level will be performed as soon as possible after the agreement as the discussion with the physician could lead to a change in dietary habits. It will be performed by high-pressure liquid chromatography (Cerba Laboratory, F-Cergy Pontoise) according to Lee et al.
2. the correlation between plasma vitamin C level and clinical signs of scurvy, especially signs of latent scurvy like tiredness, leg pain, gums involvement, previously loss of healthy teeth. These signs will be recorded in a structured questionnaire during the first consultation, before knowing the laboratory result patient. All patients who are smoking will perform systematic otorhinolaryngology examination in search of cancer. Other reasons for weakness will be searched by clinical anamneses, body examination, blood probe and abdominal ultrasound examination.
3. the decrease or disappearance of tiredness and/or purpura and/or gums involvement will be studied after vitamin C supplementation in patients whose vitamin C plasma determination is under normal levels and that don't have another explanation for their tiredness. Patients will be evaluated after receiving 1 g oral vitamin C for at least three months.

Ethical considerations The study was approved by the institutional ethics committee of the clinic and was conducted in accordance with the principles of the Declaration of Helsinki. Informed consent was obtained before entry study and each participant agreed to pay for the plasma vitamin C determination.

Dissemination findings Findings for the present study will be reported in manuscripts that will be submitted for publication to a leading medical or nutrition journal in a appropriate field (i.e.alcoholism, nutrition). In addition, findings will be presented as abstracts, posters and presentations at conferences.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteered for alcohol detoxification even if they had prior complications of excessive alcohol consumption.
* Each patient provided written consent to the study and agreed to pay himself the determination of the plasma ascorbic level.

Exclusion Criteria:

* Confusion or alcoholic coma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 51 patients volunteered to alcohol withdrawal, 14 women at a mean age of 52+/-8 (extreme 38 to 62 years) (range 24) and 37 men at a mean age of 58 +/-12 (extreme 34 to 83) (range 49).
  Three men refused the blood test and one didn't show up for the appointment. The mean age of the 33 remaining male patients was not impacted: mean age of 58 with quite the same SD (13) and the same range.
  Therefore 47 patients were included.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Plasma vitamin C concentration in alcoholic withdrawal patients | 23 months (beginning till end of the recruitment)
  Plasma vitamin C determination will be performed as soon as possible after the consent of the patient.
  Measurement of vitamin C will be performed by high-pressure liquid chromatography (Cerba Laboratory, F-Cergy Pontoise) with a Roche Fara centrifugal analyzer

SECONDARY OUTCOMES:
Correlation between plasma vitamin C and latent scurvy symptoms | 23 months (beginning till end of the recruitment)
  Using Excel, we will apply a transformation to convert status of tiredness, skin symptoms and gum involvement/ loss of healthy teeth into binary variables.This is in order to provide a better graphical representation. One graph will be displayed per symptom. When it comes to the binary variables, 0 corresponds to " absence of tiredness" whereas 1 corresponds to "presence of tiredness" for the first graph; 0 corresponds to "absence of purpura" whereas 1 means "presence of purpura " for the second graph; 0 corresponds to "absence of gums involvement or absence of loss of healthy teeth "whereas 1 means "presence of gums involvement or loss of healthy teeth".

OTHER OUTCOMES:
Questionnaire detailing the evolution of tiredness/purpura/gums involvement after supplementation with 1g/day of oral vitamin C for three months | 3 to 4 months for each patient
  Deficient or depleted patients will be supplemented with 1g/day of oral vitamin C for three months. When being examined after three months, the patients will be asked about the feeling of tiredness and the evolution of purpura and gums involvement will be investigated. Results will be expressed with binary variables (0 corresponds to a non-improvement state whereas 1 corresponds to an improvement state).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Battistelli, MD, Principal Investigator — Nouvelle Clinique des Trois Frontieres Saint-Louis

IPD SHARING:
Plan to Share IPD: Yes
Laboratory vitamin C results which will be deidentified Anonymous data displayed in an Excel table
Time Frame: Data are available immediately and till end 2019
Access Criteria: Researchers interested in alcoholism combined with nutrition

REFERENCES:
- [Background] Johnston CS, Thompson LL. Vitamin C status of an outpatient population. J Am Coll Nutr. 1998 Aug;17(4):366-70. doi: 10.1080/07315724.1998.10718777. PMID 9710847
- [Background] Hercberg S, Preziosi P, Galan P, Devanlay M, Keller H, Bourgeois C, Potier de Courcy G, Cherouvrier F. Vitamin status of a healthy French population: dietary intakes and biochemical markers. Int J Vitam Nutr Res. 1994;64(3):220-32. PMID 7814238
- [Background] Bergheim I, Parlesak A, Dierks C, Bode JC, Bode C. Nutritional deficiencies in German middle-class male alcohol consumers: relation to dietary intake and severity of liver disease. Eur J Clin Nutr. 2003 Mar;57(3):431-8. doi: 10.1038/sj.ejcn.1601557. PMID 12627180
- [Background] Lux-Battistelli C, Battistelli D. Latent scurvy with tiredness and leg pain in alcoholics: An underestimated disease three case reports. Medicine (Baltimore). 2017 Nov;96(47):e8861. doi: 10.1097/MD.0000000000008861. PMID 29382002
- [Background] Lee W, Roberts SM, Labbe RF. Ascorbic acid determination with an automated enzymatic procedure. Clin Chem. 1997 Jan;43(1):154-7. PMID 8990238
- [Background] Fain O, Paries J, Jacquart B, Le Moel G, Kettaneh A, Stirnemann J, Heron C, Sitbon M, Taleb C, Letellier E, Betari B, Gattegno L, Thomas M. Hypovitaminosis C in hospitalized patients. Eur J Intern Med. 2003 Nov;14(7):419-425. doi: 10.1016/j.ejim.2003.08.006. PMID 14614974
- [Background] Pearson JF, Pullar JM, Wilson R, Spittlehouse JK, Vissers MCM, Skidmore PML, Willis J, Cameron VA, Carr AC. Vitamin C Status Correlates with Markers of Metabolic and Cognitive Health in 50-Year-Olds: Findings of the CHALICE Cohort Study. Nutrients. 2017 Aug 3;9(8):831. doi: 10.3390/nu9080831. PMID 28771190
- [Background] Malmauret L, Leblanc J, Cuvelier I, Verger P. Dietary intakes and vitamin status of a sample of homeless people in Paris. Eur J Clin Nutr. 2002 Apr;56(4):313-20. doi: 10.1038/sj.ejcn.1601312. PMID 11965507
- [Background] Crandon JH, Lund CC, Dill DB. Experimental human scurvy. N Engl J Med 1940; 223:353-69
- [Background] Carr AC, Bozonet SM, Pullar JM, Simcock JW, Vissers MC. Human skeletal muscle ascorbate is highly responsive to changes in vitamin C intake and plasma concentrations. Am J Clin Nutr. 2013 Apr;97(4):800-7. doi: 10.3945/ajcn.112.053207. Epub 2013 Feb 27. PMID 23446899
- See also: World Health Organization: Signs and symptoms; Classic scurvy. In: Scurvy and its prevention and control in major emergencies (1999) p 4 — http://apps.who.int/iris/bitstream/10665/66962/1/WHO_NHD_99.11.pdf